CLINICAL TRIAL: NCT04971070
Title: Analysis of Related Risk Factors of Hypoglycemia Consciousness Disorder
Status: Completed | Type: Observational
Sponsor: Chongqing Renji Hospital, University of Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 31921003
Record Dates: First submitted 2021-06-23; First posted 2021-07-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-06

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoglycemic disturbance group
  Interventions: Other: Observation and follow-up
- Hypoglycemia was not a disorder of consciousness group
  Interventions: Other: Observation and follow-up

INTERVENTIONS:
Other: Observation and follow-up — Observation and follow-up study

SUMMARY:
Objective to explore the high risk factors and inducements of consciousness disorder in patients with hypoglycemia, and to conduct a retrospective study.

ELIGIBILITY:
Inclusion Criteria:

Symptoms of hypoglycemia such as palpitation, sweating and fatigue were found at the time of treatment. At the same time, the blood glucose of non-diabetic patients was less than 2.8mmol/L, and the blood glucose of diabetic patients was less than 3.9mmol/L

Exclusion Criteria:

Exclusion criteria: Although there were hypoglycemia symptoms at the time of treatment, the blood glucose of non-diabetic patients was more than 2.8mmol/L, and the blood glucose of diabetic patients was more than 3.9mmol/L.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Through retrospective control study, this study analyzed the high-risk factors and predisposing factors of hypoglycemia patients, laid a certain foundation for improving the diagnosis and treatment level of hypoglycemia consciousness disorder, and provided a certain scientific basis for further exploring the mechanism of hypoglycemia consciousness disorder
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Analysis of risk factors of hypoglycemia with disturbance of consciousness | 2021-2011
  Analysis of risk factors of hypoglycemia with disturbance of consciousness

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Renji Hospital, University of Chinese Academy of Sciences, Chongqing, Chongqing Municipality, China